CLINICAL TRIAL: NCT05774561
Title: Liquid Biopsies - a Possible Tool for Treatment Monitoring and Early Recurrence Detection in HPV-associated Diseases
Brief Title: Role of Liquid Biopsies in HPV-associated Cancer Treatment Monitoring
Status: Recruiting | Type: Observational
Sponsor: The Institute of Molecular and Translational Medicine, Czech Republic (Other)
Collaborators: National Institute for Cancer Research, Czech Republic (Other); University Hospital Olomouc (Other)
Responsible Party: Sponsor
Other Study IDs: NU-23-03-00255
Record Dates: First submitted 2023-01-24; First posted 2023-03-17 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-07

CONDITIONS: Cervical Cancer; Cervical Dysplasia; Oropharyngeal Cancer; Human Papillomavirus Infection
Keywords: human papillomavirus; HPV; liquid biopsies; cervicovaginal swab; cervical cancer; oropharyngeal cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms; Uterine Cervical Dysplasia; Oropharyngeal Neoplasms; Papillomavirus Infections | interventions — Liquid Biopsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — gargle lavage samples, oropharyngeal swabs, breath condensate, blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Arm A - Oropharyngeal cancer patients: In total, approx. 200 OPC cancer patients will be enrolled in the study Arm A, with both prospective and retrospective parts enrolling 100 OPC patients. The Arm A will enroll patients from the Department of Otorhinolaryngology and Head and Neck Surgery, University Hospital Olomouc. Pre-treatment primary samples of fresh or FFPE tissue samples will be collected. Liquid biopsies (gargle lavage, oropharyngeal smear, breath condensate, and blood sample) will be collected. Obtained samples will be tested by CE-IVD (device complies with European in vitro diagnostic Directive) marked HPV diagnostic test. A laboratory developed digital droplet PCR assay will be used for ct HPV DNA detection. Sampling will be performed at pre & post treatment check-ups, and every 3 months for 3 years and every 6 months for 2 years.
  Interventions: Diagnostic Test: Arm A - Diagnostic test: HPV detection in liquid biopsies
- Arm B - Cervical cancer patients: Into the study Arm B will be enrolled 80 patients with CC and 120 patients with HSIL, and 80 patients will be enrolled into the retrospective part. The Arm B will enroll patients from the Department of Gynecology and Obstetrics, University Hospital Olomouc. Pre-treatment primary samples of fresh or FFPE tissue samples will be collected. Liquid biopsies (cervicovaginal swab and blood sample) will be collected. Obtained samples will be tested by CE-IVD marked HPV diagnostic test. A laboratory developed digital droplet PCR assay will be used for ct HPV DNA detection. Sampling will be performed at pre & post treatment check-ups, and every 3 months for 2 years and every 6 months for 3 years.
  Interventions: Diagnostic Test: Arm B - Diagnostic test: HPV detection in liquid biopsies

INTERVENTIONS:
Diagnostic Test: Arm A - Diagnostic test: HPV detection in liquid biopsies — Patients will be asked to perform self-collection of gargle lavage samples. Oropharyngeal swabs, breath condensate, and blood samples will be taken by trained clinicians.
  Groups: Arm A - Oropharyngeal cancer patients
Diagnostic Test: Arm B - Diagnostic test: HPV detection in liquid biopsies — Patients will be asked to perform cervicovaginal self-sampling using Evalyn Brush. Blood samples will be taken by trained clinicians.
  Groups: Arm B - Cervical cancer patients

SUMMARY:
This trial will evaluate the possible benefits and the performance of liquid biopsies in HPV-associated cancer treatment monitoring. This study aims to find a combination of an adequately sensitive and specific sampling method and biomarkers for early risk stratification of disease recurrence.

DETAILED DESCRIPTION:
Although the cancers associated with human papillomavirus (HPV) infection are currently almost entirely preventable, a significant part of the Czech population suffers from these diseases. The most common HPV-associated cancers are cervical cancer (CC) and oropharyngeal cancer (OPC). In these, the severe problem is successful monitoring of the treatment effectiveness and early disease recurrence detection. It is, therefore, necessary to find a non-invasive method that could specifically and timely identify patients at risk of recurrence and thus enable patients with quality and less burdensome medical care. The use of liquid biopsies (LB), which the study focuses on, looks most promising.

This study is divided into two arms, with each arm including both prospective and retrospective parts. Into prospective parts will be enrolled only newly diagnosed CC/HSIL (high-grade cervical intraepithelial lesions) or OPC patients. In contrast, the retrospective part will enroll patients in post-treatment follow-up. In both study arms, fresh tumor tissues will be sampled from patients in prospective parts before treatment, and archived Formalin Fixed Paraffin Embedded (FFPE) tissue samples will be obtained from patients of retrospective parts.

Regarding the liquid biopsies, pre & post-treatment sampling of LB will be performed. Subsequently, regular sample acquisition will be performed during follow-up according to the standard medical practice in both prospective and retrospective parts. Oropharyngeal swabs, gargle lavage,exhaled breath condensate (EBC), and blood samples will be collected from OPC patients. Blood collection and self-sampling of cervicovaginal swabs will be performed in patients with CC/HSIL. All samples, excluding blood samples, will be tested for the presence of the most prevalent high-risk and low-risk HPV genotypes. The circulating tumor (ct) HPV DNA will be monitored in blood samples. Additionally, the mutation profile of the primary tumors will be examined in fresh and FFPE samples.

The dynamics of HPV DNA will be monitored throughout all follow-up samples and correlated with the obtained clinical data. A created panel of frequently altered genes will be used for alterations monitoring in liquid biopsies. In the final analysis of laboratory and clinical results, we assume a finding of a clinically usable algorithm that could predict the risk of disease recurrence for a particular patient.

ELIGIBILITY:
Inclusion Criteria:

Women diagnosed with CC/HSIL. Men and women diagnosed with OPC. Patients must agree with study enrollment and must sign study informed consent.

Exclusion Criteria:

No exclusion criteria are set.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Oropharyngeal cancer patients, Cervical cancer patients
Sampling Method: Non-Probability Sample
Enrollment: 480 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Dynamics of HPV infection in cervical cancer patients during 4-year follow-up. | 4 years
  HPV-status in liquid biopsies collected during pre-treatment, post-treatment and follow-up check-ups.
Dynamics of HPV infection in oropharyngeal cancer patients during 4-year follow-up. | 4 years
  HPV-status in liquid biopsies collected during pre-treatment, post-treatment and follow-up check-ups.
Dynamics of circulating tumor (ct) HPV DNA in oropharyngeal cancer patients. | 4 years
  Correlation of plasmatic ct HPV DNA level with cancer patient´s prognosis.
Dynamics of circulating tumor (ct) HPV DNA in cervical cancer patients | 4 years
  Correlation of plasmatic ct HPV DNA level with patient´s prognosis
Analysis of the mutational landscape of oropharyngeal cancer cases. | 4 years
  Correlation of tumor mutational burden (TMB) with cancer patient´s prognosis.
Analysis of the mutational landscape of cervical cancer cases. | 4 years
  Correlation of tumor mutational burden (TMB) with cancer patient´s prognosis.

CONTACTS AND LOCATIONS:
Overall Officials: Marian Hajduch, MD., PhD., Study Director — IMTM, Palacky University in Olomouc, Faculty of Medicine and Dentistry
Locations (1):
- University Hospital Olomouc, Olomouc, Czechia

IPD SHARING:
Plan to Share IPD: No